CLINICAL TRIAL: NCT03374774
Title: A Multi-centre Prospective, Non-interventional Study of Ability and Willingness to Pay for BIAsp 30 in a Real World Population With Type 2 Diabetes Mellitus
Brief Title: A Non-interventional Study of Ability and Willingness to Pay for BIAsp 30 in a Real World Population With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-4343; U1111-1195-7991 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Type 2 Diabetes Mellitus: Participants will be prescribed and treated with commercially available BIAsp 30 according to routine clinical practice at the discretion of the treating physician, independent of this study. The study will gather data over the course of routine treatment on willingness to pay for BIAsp 30 in FlexPen® or Penfill®.
  Interventions: Drug: BIAsp 30

INTERVENTIONS:
Drug: BIAsp 30 — Participants will receive commercially available BIAsp 30 according to routine clinical practice. The physician will determine the starting dose and any potential later change to the dose.

SUMMARY:
The purpose of this study is to collect information about the participant's ability and willingness to pay for NovoMix 30 using a modern device, which is prescribed to the participant by the study doctor for Type 2 Diabetes Mellitus according to routine clinical practice. The study aims to obtain data that can guide prescribers' understanding of the ability and willingness to pay for NovoMix 30 FlexPen or Penfill among participants in the growing middle class in India and Egypt. The decision to prescribe NovoMix 30 FlexPen or Penfill has been made independent from this study.

ELIGIBILITY:
Inclusion Criteria: - The decision to initiate treatment with commercially available BIAsp 30 has been made by the patient and the treating physician before and independently from the decision to include the patient in this study - Patients selected by their physician for participation in the study, who are likely to be able and willing to pay for the BIAsp 30 treatment for at least 12 weeks from baseline visit as assessed by the treating physician - Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol) - Male or female greater than or equal to 18 years at time of informed consent - Diagnosed with T2DM and treated with BHI in vials for at least three consecutive months at time of informed consent Exclusion Criteria: - Previous participation in this study. Participation is defined as having given informed consent in this study - Concurrent participation in any other clinical trial or study - Patients previously treated with insulin analogues - Known or suspected hypersensitivity to study product (or any of the excipients of the study product; a full list of excipients is provided in Summary of product characteristics (SmPC) of NovoMix® 30) or related products - Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation - Patients who are unable to read or write (illiterate)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus, previously treated with biphasic human insulin (BHI), who are prescribed and treated with commercially available BIAsp 30 from their treating physician as part of a usual care
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are using BIAsp 30 as their primary insulin | Week 12
  Proportion of patients

SECONDARY OUTCOMES:
Demographic and socio-economic characteristics of patients still using BIAsp 30 and of patients no longer using BIAsp 30 as their primary insulin, measured by Ability to Pay Questionnaire | Week 12
  This questionnaire consists of a physician's part and a patient's part. The questionnaire reflects the socio-economic and lifestyle characteristics of patients.
Change from baseline to Week 12 after first prescription of BIAsp 30 in treatment satisfaction, measured by Diabetes Treatment Satisfaction Questionnaire (status) | Week 0, week 12
  The DTSQs questionnaire will be used to assess subject's treatment satisfaction. This instrument contains 8 items and measures the treatment for your diabetes (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings regarding treatment.
Change from baseline to Week 12 after first prescription of BIAsp 30 in patient evaluation of delivery system, measured by Treatment Related Impact Measure for Diabetes (TRIM-D) Device | Week 0, week 12
  The TRIM-D Device is an eight item measure with two domains assessing Device Bother and Device Function. This captures information on the ease of use, convenience, and handling of the device(s) used to take diabetes medication. The measure has acceptable reliability, validity and ability to detect change.
Diabetes Pen Experience Measure (DPEM) Scores (proportions of each item) | Week 0
  This measure captures information on the convenience, user friendliness, and handling of pen, which is used to administer BIAsp 30. Seven items are scored on a 5 point scale from 'Not at all' to 'Extremely'. Proportion of each item to be presented.
Weighted patient preferences for treatment attributes derived from the Discrete Choice Experiment (DCE) | Week 0
  Through multiple scenarios, each patient will be prompted to select the choice that seems most favourable to the patient. Each scenario will consist of a bundled collection of attributes relevant for insulin therapy. The questionnaire consists of approximately nine questions/scenarios for each patient.
Diabetes Pen Experience Measure (DPEM) Scores (frequency of each item) | Week 0
  This measure captures information on the convenience, user friendliness, and handling of pen, which is used to administer BIAsp 30. Seven items are scored on a 5 point scale from 'Not at all' to 'Extremely'. Frequency of each item to be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (15):
- India (15):
  - Novo Nordisk Investigational Site, Guwahati, Assam
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kalaburagi, Karnataka
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Kolhāpur, Maharashtra
  - Novo Nordisk Investigational Site, Nashik, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Lucknow, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Belagavi
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Thriruvananthapuram

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Murthy S, Aneja P, Asirvatham AJ, Husemoen LLN, Rhee NA, Kesavadev J. Understanding Patients' Willingness to Pay for Biphasic Insulin Aspart 30/70 in a Pen Device for Type 2 Diabetes Treatment in an Out-of-Pocket Payment Market. Pharmacoecon Open. 2021 Jun;5(2):261-273. doi: 10.1007/s41669-020-00246-3. Epub 2021 Jan 6. PMID 33410093